CLINICAL TRIAL: NCT02639052
Title: Itch Relieving Effect of Botox: a Study in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23230; 126938 (Other: FDA IND)
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Pruritus
Keywords: Itch; Botox; Healthy Volunteers
MeSH Terms: conditions — Pruritus | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Experimental): 10 units of Botox intradermally injected into one forearm. The subject is blinded to which forearm receives the Botox and which forearm receives the saline vehicle.
  Interventions: Drug: Botox
- Saline (Placebo Comparator): Saline vehicle intradermally injected into the other forearm. The subject is blinded to which forearm receives the Botox and which forearm receives the saline vehicle.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botox — 10 units of Botox will be intradermally injected into one 4x4cm area on the volar forearm on 1st study visit.
  Arms: Botox
Drug: Saline — 10 units of the Saline vehicle will be intradermally injected into one 4x4cm area on the contralateral volar forearm on the 1st study visit.
  Arms: Saline

SUMMARY:
The purpose of this study is to determine if Botox is effective in the treatment of an experimentally induced itch that mimics chronic itch in healthy volunteers.

DETAILED DESCRIPTION:
Several studies have shown that botulinum toxin type A (BoNT/A) has an antipruritic effect due to the inhibition of acetylcholine and other pruritic factors, such as substance P and glutamate. For instance, subcutaneous BoNT/A improves itch accompanied to hand eczema, dermatitis, lichen simplex, and rhinitis. Furthermore, a double-blind, placebo-controlled study showed that BoNT/A reduced histamine itch intensity in healthy men. Since acetylcholine has been shown to mediate itch in atopic dermatitis, this study aims to test the itch relieving effect of BoNT/A on a non-histaminergic model for chronic itch. This non-histaminergic model using the plant cowhage induces itch by activating protease activated receptor 2 (PAR2) receptors, which play a role in the itch of atopic dermatitis, also making this model better suited to test the efficacy of BoNT/A to relive chronic itch.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers between 18 and 50 years of age.
2. Must be in general good health with no disease or physical conditions that would impair evaluation of itch and pain perception.
3. No history of chronic itch or pain.
4. Must abstain from the use of any systemic or topical anti-histamine, steroid, or pain relief medications from the week prior to the study till the completion of the study.
5. Must abstain from the use of moisturizers on the arm.

Exclusion Criteria:

1. Individuals under 18 or over 50 years of age.
2. Inability to complete the required measures.
3. The presence of an itchy skin disease.
4. Diagnosis of diseased that would affect itch or pain perception (e.g. neuropathies).
5. Currently enrolled in any investigational study in which the subject is receiving any type of drug, biological, or non-drug therapy.
6. Use of oral, topical analgesics, or other medications known to interfere with itch or pain perception in the week prior to the study and throughout the study (e.g. antihistamines, anesthetics, opioids, neuroleptics, etc.).
7. Use of emollients on the arms a week prior to the study and throughout the study.
8. Use of anti-depressants, anti-psychotics, and illicit drugs.
9. Known history of neuropathy, uremia, uncontrolled thyroid disease, and diabetes mellitus.
10. Use of Botulinum toxin in the last year.
11. Known allergies to Botox.
12. Pregnant women. (Women of child bearing potential will undergo an human chorionic gonadotrophin (hCG) pregnancy test before Botox application).
13. Hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation.
14. Infection at the injection site.
15. Cardiovascular disease.
16. Neuromuscular disorder (e.g., amyotrophic lateral sclerosis, myasthenia gravis, or Lambert-Eaton syndrome).
17. Compromised respiratory function.
18. Dysphagia.
19. History of urinary tract infection.
20. History of urinary retention.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Temple University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang W, Foster JA, Rogachefsky AS. Pharmacology of botulinum toxin. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):249-59. doi: 10.1067/mjd.2000.105567. PMID 10906647
- [Background] Hallett M. How does botulinum toxin work? Ann Neurol. 2000 Jul;48(1):7-8. No abstract available. PMID 10894209
- [Background] Ishikawa H, Mitsui Y, Yoshitomi T, Mashimo K, Aoki S, Mukuno K, Shimizu K. Presynaptic effects of botulinum toxin type A on the neuronally evoked response of albino and pigmented rabbit iris sphincter and dilator muscles. Jpn J Ophthalmol. 2000 Mar-Apr;44(2):106-9. doi: 10.1016/s0021-5155(99)00197-5. PMID 10715374
- [Background] Cui M, Khanijou S, Rubino J, Aoki KR. Subcutaneous administration of botulinum toxin A reduces formalin-induced pain. Pain. 2004 Jan;107(1-2):125-33. doi: 10.1016/j.pain.2003.10.008. PMID 14715398
- [Background] Wollina U, Karamfilov T. Adjuvant botulinum toxin A in dyshidrotic hand eczema: a controlled prospective pilot study with left-right comparison. J Eur Acad Dermatol Venereol. 2002 Jan;16(1):40-2. doi: 10.1046/j.1468-3083.2002.00361.x. PMID 11952288
- [Background] Swartling C, Naver H, Lindberg M, Anveden I. Treatment of dyshidrotic hand dermatitis with intradermal botulinum toxin. J Am Acad Dermatol. 2002 Nov;47(5):667-71. doi: 10.1067/mjd.2002.124605. PMID 12399757
- [Background] Heckmann M, Heyer G, Brunner B, Plewig G. Botulinum toxin type A injection in the treatment of lichen simplex: an open pilot study. J Am Acad Dermatol. 2002 Apr;46(4):617-9. doi: 10.1067/mjd.2002.120455. PMID 11907521
- [Background] Unal M, Sevim S, Dogu O, Vayisoglu Y, Kanik A. Effect of botulinum toxin type A on nasal symptoms in patients with allergic rhinitis: a double-blind, placebo-controlled clinical trial. Acta Otolaryngol. 2003 Dec;123(9):1060-3. doi: 10.1080/00016480310000755. PMID 14710908
- [Background] Gazerani P, Pedersen NS, Drewes AM, Arendt-Nielsen L. Botulinum toxin type A reduces histamine-induced itch and vasomotor responses in human skin. Br J Dermatol. 2009 Oct;161(4):737-45. doi: 10.1111/j.1365-2133.2009.09305.x. Epub 2009 May 11. PMID 19624547
- [Background] Heyer G, Vogelgsang M, Hornstein OP. Acetylcholine is an inducer of itching in patients with atopic eczema. J Dermatol. 1997 Oct;24(10):621-5. doi: 10.1111/j.1346-8138.1997.tb02305.x. PMID 9375459
- [Background] Wessler I, Reinheimer T, Kilbinger H, Bittinger F, Kirkpatrick CJ, Saloga J, Knop J. Increased acetylcholine levels in skin biopsies of patients with atopic dermatitis. Life Sci. 2003 Mar 28;72(18-19):2169-72. doi: 10.1016/s0024-3205(03)00079-1. PMID 12628475
- [Background] Reddy VB, Iuga AO, Shimada SG, LaMotte RH, Lerner EA. Cowhage-evoked itch is mediated by a novel cysteine protease: a ligand of protease-activated receptors. J Neurosci. 2008 Apr 23;28(17):4331-5. doi: 10.1523/JNEUROSCI.0716-08.2008. PMID 18434511
- [Background] Papoiu AD, Tey HL, Coghill RC, Wang H, Yosipovitch G. Cowhage-induced itch as an experimental model for pruritus. A comparative study with histamine-induced itch. PLoS One. 2011 Mar 14;6(3):e17786. doi: 10.1371/journal.pone.0017786. PMID 21423808

RESULTS

PARTICIPANT FLOW:
Groups:
- Botox and Saline Vehicle Control: 10 units of both Botox and a saline vehicle will be intradermally injected into one forearm or the other on the first study visit. The subject will be blinded to which forearm receives the Botox and which forearm receives the saline vehicle.
  Botox: 10 units of Botox will be intradermally injected into one 4x4cm area on the volar forearm on 1st study visit.
  Saline: 10 units of the Saline vehicle will be intradermally injected into one 4x4cm area on the contralateral volar forearm on the 1st study visit.
Period: Overall Study
Arm/Group | Botox and Saline Vehicle Control
Started | 35
Visit 1 (Baseline) | 35
Visit 2 (1-week Follow-up) | 35
Visit 3 (1-month Follow-up) | 35
Visit 4 (3-month Follow-up) | 34
Completed | 34
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Botox and Saline Vehicle Control
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Itch by VAS Itch Intensity at Baseline (Visit 1)
Description: The primary endpoint is to test the antipruritic effect of Botox using an itch visual analog scale (VAS) intensity scale as an outcome measure. The itch VAS intensity scale ranges from a minimum of 0 (no itch - best) to a maximum of 10 (maximum itch - worst). Participants will rate itch intensity after itch is induced with cowhage.
Time Frame: Baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox: 10 units of Botox intradermally injected into one forearm
- Saline: Saline vehicle intradermally injected into the other forearm
Arm/Group | Botox | Saline
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline (Visit 1), 0 seconds | 4.5 (2.8) | 4.3 (2.8)
  Baseline (Visit 1), 30 seconds | 6.5 (2.6) | 6.3 (2.3)
  Baseline (Visit 1), 60 seconds | 6.8 (2.2) | 6.5 (2.1)
  Baseline (Visit 1), 90 seconds | 5.9 (2.1) | 6.3 (1.5)
  Baseline (Visit 1), 120 seconds | 5.1 (2.2) | 5.1 (2.0)
  Baseline (Visit 1), 150 seconds | 4.1 (2.2) | 3.9 (2.1)
  Baseline (Visit 1), 180 seconds | 2.8 (2.0) | 2.8 (1.8)
  Baseline (Visit 1), 210 seconds | 2.0 (1.6) | 2.0 (1.8)
  Baseline (Visit 1), 240 seconds | 1.3 (1.5) | 1.4 (1.7)
  Baseline (Visit 1), 270 seconds | 0.9 (1.3) | 0.9 (1.6)
  Baseline (Visit 1), 300 seconds | 0.6 (1.1) | 0.9 (1.5)
  Baseline (Visit 1), All Times | 3.7 (3.0) | 3.7 (2.9)
Statistical Analysis 1: Comparison: Botox vs Saline; Baseline assessment of itch VAS after itch induction but prior to Botox or saline application. Analyzed using ANOVA with repeated measures to compare main effects of treatment (Botox vs saline) and time, and interaction effect between treatment and time; Test type: Superiority or Other; p = 0.9704, ANOVA with Repeated Measures — Significance defined a priori as p<0.05. P-values not adjusted for multiple comparisons

2. Primary Outcome: Itch by VAS Itch Intensity at 1 Week (Visit 2)
Description: as for outcome 1
Time Frame: 1 week from Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Saline
Number analyzed (Participants) | 35 | 35
units on a scale
  1 Week (Visit 2), 0 seconds | 3.3 (2.4) | 4.0 (2.9)
  1 Week (Visit 2), 30 seconds | 5.4 (2.3) | 6.7 (2.2)
  1 Week (Visit 2), 60 seconds | 5.9 (2.3) | 6.9 (2.1)
  1 Week (Visit 2), 90 seconds | 4.9 (2.3) | 6.1 (1.7)
  1 Week (Visit 2), 120 seconds | 3.7 (2.4) | 4.8 (2.0)
  1 Week (Visit 2), 150 seconds | 2.7 (2.5) | 3.8 (2.2)
  1 Week (Visit 2), 180 seconds | 2.0 (2.3) | 2.7 (2.1)
  1 Week (Visit 2), 210 seconds | 1.4 (1.8) | 1.9 (1.9)
  1 Week (Visit 2), 240 seconds | 0.9 (1.5) | 1.3 (1.6)
  1 Week (Visit 2), 270 seconds | 0.6 (1.3) | 0.9 (1.3)
  1 Week (Visit 2), 300 seconds | 0.4 (1.1) | 0.7 (1.3)
  1 Week (Visit 2), All Times | 2.8 (2.8) | 3.6 (2.9)
Statistical Analysis 1: Comparison: Botox vs Saline; 1 week (Visit 2) was the first assessment of itch VAS after itch induction after Botox or saline application. Analyzed using ANOVA with repeated measures to compare main effects of treatment (Botox vs saline) and time, and interaction effect between treatment and time; Test type: Superiority or Other; p < 0.0001, ANOVA with Repeated Measures — Statistical significance defined a priori as p<0.05. P-values have not been adjusted for multiple comparisons

3. Primary Outcome: Itch by VAS Itch Intensity at 1 Month (Visit 3)
Description: as for outcome 1
Time Frame: 1 Month from Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Saline
Number analyzed (Participants) | 35 | 35
units on a scale
  1 Month (Visit 3), 0 seconds | 3.2 (2.6) | 3.8 (2.8)
  1 Month (Visit 3), 30 seconds | 5.0 (2.6) | 6.2 (2.4)
  1 Month (Visit 3), 60 seconds | 5.1 (2.3) | 6.2 (1.8)
  1 Month (Visit 3), 90 seconds | 4.3 (2.3) | 5.7 (2.3)
  1 Month (Visit 3), 120 seconds | 3.5 (2.0) | 4.5 (2.4)
  1 Month (Visit 3), 150 seconds | 2.3 (1.8) | 3.3 (2.2)
  1 Month (Visit 3), 180 seconds | 1.5 (1.4) | 2.2 (2.1)
  1 Month (Visit 3), 210 seconds | 0.9 (1.3) | 1.4 (1.7)
  1 Month (Visit 3), 240 seconds | 0.7 (1.0) | 0.9 (1.3)
  1 Month (Visit 3), 270 seconds | 0.3 (0.7) | 0.6 (1.0)
  1 Month (Visit 3), 300 seconds | 0.2 (0.5) | 0.4 (0.8)
  1 Month (Visit 3), All Times | 2.5 (2.5) | 3.2 (2.9)
Statistical Analysis 1: Comparison: Botox vs Saline; 1 month (Visit 3) was the second assessment of itch VAS after itch induction after Botox or saline application. Analyzed using ANOVA with repeated measures to compare main effects of treatment (Botox vs saline) and time, and interaction effect between treatment and time; Test type: Superiority or Other; p < 0.0001, ANOVA with Repeated Measures — Statistically significant difference in mean itch VAS between the two treatments (Botox mean=2.45 versus saline mean=3.20, p<0.0001). Statistical significance defined a priori as p<0.05. P-values have not been adjusted for multiple comparisons

4. Primary Outcome: Itch by VAS Itch Intensity at 3 Months (Visit 4)
Description: as for outcome 1
Time Frame: 3 Months from Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Saline
Number analyzed (Participants) | 34 | 34
units on a scale
  3 Months (Visit 4), 0 seconds | 2.3 (1.8) | 3.3 (2.4)
  3 Months (Visit 4), 30 seconds | 4.5 (2.5) | 5.4 (2.5)
  3 Months (Visit 4), 60 seconds | 4.9 (2.3) | 5.9 (2.2)
  3 Months (Visit 4), 90 seconds | 4.6 (2.3) | 5.2 (2.1)
  3 Months (Visit 4), 120 seconds | 3.8 (2.0) | 4.7 (2.1)
  3 Months (Visit 4), 150 seconds | 3.0 (2.0) | 3.6 (2.1)
  3 Months (Visit 4), 180 seconds | 2.1 (1.9) | 2.8 (1.9)
  3 Months (Visit 4), 210 seconds | 1.5 (1.7) | 1.9 (1.9)
  3 Months (Visit 4), 240 seconds | 1.0 (1.2) | 1.4 (1.6)
  3 Months (Visit 4), 270 seconds | 0.7 (1.1) | 0.9 (1.4)
  3 Months (Visit 4), 300 seconds | 0.3 (0.6) | 0.6 (1.1)
  3 Months (Visit 4), All Times | 2.6 (2.4) | 3.2 (2.7)
Statistical Analysis 1: Comparison: Botox vs Saline; 3 months (Visit 4) was the third assessment of itch VAS after itch induction after Botox or saline application. Analyzed using ANOVA with repeated measures to compare main effects of treatment (Botox vs saline) and time, and interaction effect between treatment and time; Test type: Superiority or Other; p = 0.0004, ANOVA with Repeated Measures — Statistical significance defined a priori as p<0.05. P-values have not been adjusted for multiple comparisons; Analyzed using ANOVA with repeated measures to compare treatment (Botox vs saline), time, and interaction effect between treatment & time

5. Secondary Outcome: Change in Heat Pain Relief by VAS Pain Intensity Reporting After 1 Week, 1 Month, and 3 Months After Treatment
Description: A secondary endpoint is to see if Botox has a relieving effect on heat pain using a pain visual analog scale (VAS) intensity scale as an outcome measure. The pain VAS intensity scale ranges from a minimum of 0 (no pain - best) to a maximum of 10 (maximum pain - worst). Participants will rate pain intensity after pain is induced with a heat thermode.
Time Frame: Baseline, 1 week, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Saline
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline | 3.6 (2.4) | 3.7 (2.2)
  1 Week | 3.7 (2.5) | 3.7 (2.5)
  1 Month | 3.7 (2.5) | 4.1 (2.6)
  3 Months | 4.1 (2.4) | 4.3 (2.5)
  All Visits | 3.8 (2.4) | 4.0 (2.4)
Statistical Analysis 1: Comparison: Botox vs Saline; Analyzed using ANOVA with repeated measures to compare main effects of treatment (Botox vs saline) and visit, and interaction effect between treatment and visit; Test type: Superiority or Other; p = 0.1306, ANOVA with Repeated Measures — Statistical significance defined a priori as p<0.05

ADVERSE EVENTS:
Time Frame: Baseline, 1 week, 1 month, 3 months
Arm/Group | Botox | Saline
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes